CLINICAL TRIAL: NCT04323150
Title: The Effect of Closed Suction System on the Incidence of Ventilator-associated Pneumonia, Respiratory-associated Microbiome and Contamination of Inanimate Surfaces: a Pilot Study.
Brief Title: The Effect of Closed Suction System on the Incidence of Ventilator-associated Pneumonia.
Acronym: CSS-VAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northern State Medical University (Other)
Responsible Party: Principal Investigator, Vsevolod V. Kuzkov, Professor of the Department of Anaesthesiology and Intensive Care Medicine, MD, PhD, Northern State Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CSS-VAP-1
Record Dates: First submitted 2020-03-21; First posted 2020-03-26 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-04

CONDITIONS: Severe Traumatic Brain Injury; Pancreatic Diseases; Trauma Injury; Seizures; Encephalitis; Abdominal Sepsis
MeSH Terms: conditions — Brain Injuries, Traumatic; Pancreatic Diseases; Accidental Injuries; Seizures; Encephalitis; Intraabdominal Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Closed suction systems (Experimental)
  Interventions: Device: Closed suction systems
- Open (conventional) suction (Other): control group
  Interventions: Device: Conventional suction system

INTERVENTIONS:
Device: Closed suction systems — Closed suction systems are using for prevention of the ventilator-associated pneumoniae
  Arms: Closed suction systems
Device: Conventional suction system — The using of open (conventional) suctioning
  Arms: Open (conventional) suction

SUMMARY:
The investigators are suggesting that closed suction systems may reduce the risk of the ventilator - associated pneumoniae (VAP) and the contamination of the closest unanimated surfaces. In 2011 David et al. have shown that closed suction systems might reduce the incidence of the late VAP. Research team is thinking that preventive bundle with closed suction systems can prevent to onset of the VAP. All enrolled patients is randomizing into two groups: control group - conventional suctioning and research group - suctioning with closed suction system.

ELIGIBILITY:
Inclusion Criteria:

* invasive mechanical ventilation beyond 48 hours

Exclusion Criteria:

* hospital - acquired pneumonia
* community - acquired pneumoniae
* BMI > 35 kg/cm2
* pregnancy
* tracheostomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
incidence of the ventilator - associated pneumoniae (VAP) | Change from Baseline CPIS at 96 hours
  Assessment of CPIS, if CPIS equal or more 6 points VAP will be observed
Contamination of closet inanimate surfaces | Change from Baseline Microbiology researching at 96 hours
  Microbiology researching samples from circuit of a respirator and a bed

SECONDARY OUTCOMES:
Organ dysfunction | Change from Baseline SOFA at 96 hours
  Patient examination with Sequential Organ Function Assessment (SOFA)
Mortality | 28 days
  Mortality for 28 days of a hospitalization
C - reactive protein | Change from Baseline CRP researching at 96 hours
  Investigation of a Biomarker of the VAP
Procalcitonin | Change from Baseline CRP researching at 96 hours
  Investigation of a Biomarker of the VAP
sTREM 1 | Change from Baseline CRP researching at 96 hours
  Investigation of a Biomarker of the VAP

CONTACTS AND LOCATIONS:
Locations (1):
- State Budgetary Healthcare Institution of Arkhangelsk Region "Severodvinsk City Clinical Emergency Hospital # 2", Severodvinsk, Russia

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol